CLINICAL TRIAL: NCT02258815
Title: Phase II Feasability Study Using ch14.18/CHO Antibody and Subcutaneous Interleukin 2 After Haploidentical Stem Cell Transplantation in Children With Relapsed Neuroblastoma
Brief Title: CH14.18 1021 Antibody and IL2 After Haplo SCT in Children With Relapsed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Children's Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Peter Lang, Head of stem cell transplantation unit, University Children's Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT:2009-015936-14
Record Dates: First submitted 2013-08-07; First posted 2014-10-07 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Neuroblastoma Recurrent
Keywords: pediatric; haploidentical; stem cell transplantation
MeSH Terms: interventions — dinutuximab; humanized 3F8 anti-GD2 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ch14.18 (Experimental): A six courses regimen consisting of a 8 hour infusion (ch14.18/CHOmAb 20 mg/m² ) for five consecutive days will be administered every 4 weeks.
  Interleukin 2 will be added to cycles 4-6 at days 6,8,10 (1 x 106 IU/m²/d s.c.) Participants will be premedicated with an intravenous antihistamine and ranitidine within approximately 30 minutes prior and during the infusion of the study agent Pain as an anticipated side effect is managed by a standard pain prophylaxis with Morphium hydrochloride Disease status will be evaluated after 3 and 6 courses and after 1 year.
  Interventions: Drug: ch14.18/CHO

INTERVENTIONS:
Drug: ch14.18/CHO — A six courses regimen consisting of a 8 hour infusion (ch14.18/CHOmAb 20 mg/m² ) for five consecutive days will be administered every 4 weeks.
  Interleukin 2 will be added to cycles 4-6 at days 6,8,10 (1 x 106 IU/m²/d s.c.) Participants will be premedicated with an intravenous antihistamine and ranitidine within approximately 30 minutes prior and during the infusion of the study agent Pain as an anticipated side effect is managed by a standard pain prophylaxis with Morphium hydrochloride Disease status will be evaluated after 3 and 6 courses and after 1 year.
  Other Names: ch14.18; anti GD2 antibody

SUMMARY:
A six courses regimen consisting of a 8 hour infusion (ch14.18/CHOmAb 20 mg/m²) for five consecutive days will be administered every 4 weeks, starting 60-180 days after previous haploidentical stem cell transplantation.

Interleukin 2 will be added to cycles 4-6 at days 6,8,10 (1 x 106 IU/m²/d s.c.) Participants will be premedicated with an intravenous antihistamine and ranitidine within approximately 30 minutes prior and during the infusion of the study agent Pain as an anticipated side effect is managed by a standard pain prophylaxis with Morphium hydrochloride Disease status will be evaluated after 3 and 6 courses and after 1 year

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 21 years of age.
* Histologically confirmed neuroblastoma.
* Refractory to standard treatment (i.e. refractory disease) or relapse after previous autologous or allogenic stem cell transplantation.
* Patient has undergone haploidentical stem cell transplantation prior to antibody infusion according to appendix IV at least 60 days prior to starting immunotherapy.
* Serum glutamate pyruvate transaminase (SGPT) less than 2.5 times the upper limit of normal for age and total bilirubin less than 2 times the upper limit of normal for age. D-Dimers less than 2 times the upper limit of normal.

Creatinine clearance or radioisotope GFR greater than or equal to 40 ml/min/1.73m2.

* Cardiac shortening fraction greater than or equal to 20% by echocardiogram. Karnofsky/Lansky performance score (age appropriate) of greater than or equal to 50.
* Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
* Written informed consent is obtained, and for minors a written agreement by parents or legal guardian.

Exclusion Criteria:

* Marked baseline prolongation of QT/QTc interval (e.g. demonstration of a QTc interval > 450 milliseconds).
* Patients with symptoms of congestive heart failure or uncontrolled cardiac rhythm disturbance.
* Patients with significant psychiatric disabilities or uncontrolled seizure disorders.
* Patients with active infections or active peptic ulcer, unless these conditions are corrected or controlled.
* Patients with acute GvHD Grade III or IV or extensive chronic GvHD.
* Patients with clinically significant, symptomatic, pleural effusions.
* Patients who have had major surgery, (i.e. laparotomy or thoracotomy) within the past two weeks.
* Patients who will more than 12 months post haploidentical stem cell transplantation at the time of starting the first cycle of immunotherapy.
* Prior administration of ch14.18 antibody after allogeneic stem cell transplantation (prior administration after autologous transplantation will be acceptable)
* HIV or Hepatitis B Surface (HBS) Ag positive. As presence of either may influence the ability if the immune system to be stimulated by this treatment.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Success of treatment | 180 days
  Primary endpoint is "success of treatment" defined as a patient receiving the full protocol treatment, still alive 180 days after treatment without progression and without unacceptable toxicity and acute GvHD >= Grade III or extensive chronic GvHD.
  Thus, a composite variable is used as primary endpoint: Treatment success, is defined as a patients who did not experience
  1. unacceptable toxicities
  2. acute GvHD >= Grade III or extensive chronic GvHD
  3. other toxicities that did not recover to <= Grade 1 within 4 weeks or
  4. progressive disease after 6 cycles or
  5. deaths within treatment after SCT
  6. withdrawal due to other reasons

SECONDARY OUTCOMES:
Anti tumour responses | 1 year
  • To evaluate the anti-tumour responses resulting from this immunotherapy regimen through clinical assessments (radiographic and clinical measurements, including bone marrow immunohistochemistry for those research participants with marrow involvement).
Pharmakoinetics | 1 Year
  * To evaluate pharmacokinetics of the ch14.18/CHO including analysis of cytokine levels in patients blood during administration. Antibody levels will be evaluated in determined intervals during Therapy
NK Cell aktivation and proliferation | 1 Year
  * To evaluate changes in NK cell activation and proliferation (immunological monitoring) for additional support of potential Anti-tumor effect.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lang, MD, PhD, Principal Investigator — University Hospital Tuebingen
Locations (4):
- Austria (2):
  - University Hospital Graz, Graz
  - St. Anna Childrens Hospital, Vienna
- Germany (2):
  - University Hospital Greifswald, Greifswald
  - University Hospital Tuebingen, Tübingen

REFERENCES:
- [Derived] Flaadt T, Ladenstein RL, Ebinger M, Lode HN, Arnardottir HB, Poetschger U, Schwinger W, Meisel R, Schuster FR, Doring M, Ambros PF, Queudeville M, Fuchs J, Warmann SW, Schafer J, Seitz C, Schlegel P, Brecht IB, Holzer U, Feuchtinger T, Simon T, Schulte JH, Eggert A, Teltschik HM, Illhardt T, Handgretinger R, Lang P. Anti-GD2 Antibody Dinutuximab Beta and Low-Dose Interleukin 2 After Haploidentical Stem-Cell Transplantation in Patients With Relapsed Neuroblastoma: A Multicenter, Phase I/II Trial. J Clin Oncol. 2023 Jun 10;41(17):3135-3148. doi: 10.1200/JCO.22.01630. Epub 2023 Feb 28. PMID 36854071
- [Derived] Seitz CM, Flaadt T, Mezger M, Lang AM, Michaelis S, Katz M, Syring D, Joechner A, Rabsteyn A, Siebert N, Troschke-Meurer S, Zumpe M, Lode HN, Yang SF, Atar D, Mast AS, Scheuermann S, Heubach F, Handgretinger R, Lang P, Schlegel P. Immunomonitoring of Stage IV Relapsed Neuroblastoma Patients Undergoing Haploidentical Hematopoietic Stem Cell Transplantation and Subsequent GD2 (ch14.18/CHO) Antibody Treatment. Front Immunol. 2021 Jul 22;12:690467. doi: 10.3389/fimmu.2021.690467. eCollection 2021. PMID 34367149